CLINICAL TRIAL: NCT05027061
Title: Retrospective Medical Chart Review Study for Non-valvular Atrial Fibrillation Patients Treated or Untreated With Oral Anticoagulant in the National Cerebral and Cardiovascular Center (NCVC) in Japan
Brief Title: A Study of Participants With Non-Valvular Atrial Fibrillation (NVAF) Treated or Untreated With Oral Anticoagulant in the National Cerebral and Cardiovascular Center (NCVC) in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-771
Record Dates: First submitted 2021-08-26; First posted 2021-08-30 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Non-Valvular Atrial Fibrillation (NVAF)
Keywords: BMS-562247; Apixaban; Atrial fibrillation; Oral Anticoagulants; Japan; Retrospective Study
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Cohort 1: Non-valvular atrial fibrillation (NVAF) participants receiving oral anticoagulant - Warfarin
- Cohort 2: NVAF participants receiving oral anticoagulant - Apixaban
- Cohort 3: NVAF participants receiving oral anticoagulant - Dabigatran
- Cohort 4: NVAF participants receiving oral anticoagulant - Edoxaban
- Cohort 5: NVAF participants receiving oral anticoagulant - Rivaroxaban
- Cohort 6: NVAF participants not receiving oral anticoagulants

SUMMARY:
The purpose of this observational study is to understand real-world oral anticoagulants (OAC) (warfarin, apixaban, dabigatran, edoxaban and rivaroxaban) usage for non-valvular atrial fibrillation (NVAF) patients.

ELIGIBILITY:
Inclusion Criteria:

• Participants received medical treatment for NVAF between 10-Jan-2012 and 31-Aug-2020.

Exclusion Criteria:

* Had no data of serum creatinine in the participant's medical records
* Had no data of body weight in the participant's medical records
* Were given oral anticoagulant (OAC) for treatment of diseases other than atrial fibrillation (AF)

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of an estimated 12,000 Non-valvular atrial fibrillation (NVAF) participants' medical charts that will fulfill the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 11776 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Specialization of the treating physician | At Baseline
Distribution of socio-demographic characteristics of NVAF participants: Age group | At Baseline
Distribution of socio-demographic characteristics of NVAF participants: Gender | At Baseline
Distribution of socio-demographic characteristics of NVAF participants: Body weight | At Baseline
Distribution of socio-demographic characteristics of NVAF participants: Height | At Baseline
Distribution of socio-demographic characteristics of NVAF participants: Body mass index (BMI) | At Baseline
Distribution of outcomes of NVAF participants: Drinking information | At Baseline
Distribution of outcomes of NVAF participants: Smoking information | At Baseline
Distribution of outcomes of NVAF participants: Internal medical device information | At Baseline
Distribution of outcomes of NVAF participants: Degree of life freedom | At Baseline
Distribution of outcomes of NVAF participants: Hospitalization/outpatient status | At Baseline
Distribution of outcomes of NVAF participants: Systolic and diastolic blood pressure | At Baseline
Distribution of outcomes of NVAF participants: Pulse rate | At Baseline
Distribution of clinical characteristics of NVAF participants: Risk factors for stroke | At Baseline
Distribution of clinical characteristics of NVAF participants: Risk factors for bleeding | At Baseline
Distribution of clinical characteristics of NVAF participants: Comorbidities | At Baseline
Distribution of outcomes of NVAF participants: OAC prescription and administration status | At Baseline
Distribution of medication prescribed during baseline: angiotensin-converting enzyme inhibitor (ACE) | At Baseline
Distribution of medication prescribed during baseline: angiotensin-receptor blocker (ARB) | At Baseline
Distribution of medication prescribed during baseline: calcium antagonist | At Baseline
Distribution of medication prescribed during baseline: Antiarrhythmic drug | At Baseline
Distribution of medication prescribed during baseline: Statin | At Baseline
Distribution of medication prescribed during baseline: proton pump inhibitor (PPI) | At Baseline
Distribution of medication prescribed during baseline: H2-receptor antagonist | At Baseline
Distribution of medication prescribed during baseline: aspirin | At Baseline
Distribution of medication prescribed during baseline: P2Y12 inhibitor | At Baseline
Distribution of medication prescribed during baseline: Other antiplatelet drugs | At Baseline
Distribution of medication prescribed during baseline: Other anticoagulants | At Baseline
Distribution of medication prescribed during baseline: P-glycoprotein inhibitor | At Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm